CLINICAL TRIAL: NCT03997656
Title: A Randomised Controlled Trial of a Digital Therapy for Diabetes Prevention
Brief Title: A Digital Therapy for Diabetes Prevention Among Overweight Adults in Terengganu, Malaysia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sultan Zainal Abidin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/77
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pre Diabetes; Overweight and Obesity
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Control group
Who Masked: Investigator
Masking Description: Single-blinded approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyDipp (Experimental): The participants will go through 16-weekly core lessons that need to be completed within the first 24 weeks after randomisation focusing on changing dietary habits, increase physical activity and relapse prevention and 6-monthly post-core lessons focusing on maintenance of lifestyle habits and weight loss achieved during the core program. Each lesson will take 30 to 60 minutes to complete. The lesson will be considered complete if the participants clicked through all of the pages and answered multiple choice questions to indicate engagement and understanding.
  Interventions: Behavioral: MyDiPP (Malaysia Diabetes Prevention Program)
- Control (Other): Participants in the control group (usual care) will receive standard health education from primary care providers in the clinic. In addition, they also will be provided with pamphlets and booklets about various health topics. They will be given a diary to record their weights, diet, physical activities and blood test result.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: MyDiPP (Malaysia Diabetes Prevention Program) — The participants will go through 16-weekly core lessons that need to be completed within the first 24 weeks after randomisation focusing on changing dietary habits, increase physical activity and relapse prevention and 6-monthly post-core lessons focusing on maintenance of lifestyle habits and weight loss achieved during the core program.
  Arms: MyDipp
Other: usual care — standard health education from primary care providers in the clinic
  Arms: Control

SUMMARY:
The modern world revolves around technology; unsurprisingly companies are leveraging the expertise of the digital tech industry to aid in the prevention of chronic diseases. Among one of the most common chronic diseases in Malaysia is diabetes. Prevalence of diabetes in Malaysia has increased by more than two folds over the past two decades. Despite a growing number of tech products developments on diabetes prevention, a recent meta-analysis has found almost no evidence on digital therapy outside the developed world. Therefore, this study is needed to demonstrate the potential of digital therapy in preventing diabetes in Malaysia. The study design is a randomized controlled trial study conducted in Kuala Terengganu, Malaysia. The study will be conducted in two phases. The first phase will involve preparation of intervention modules and development of intervention mobile app. The second phase will involve validation and utilization of the digital therapy. We hope that this digital therapy program can make a significant difference in health outcomes, especially for diabetes. By giving precise regimes and daily monitoring, digital therapeutics can offer mountains of data that can potentially provide doctors unprecedented insights into patient behavior and create feedback or optimization loops for individual patients. Enabling patients to take greater control over managing their chronic illnesses and preventing disease progression could save billions of ringgits throughout the entire Malaysia healthcare system. By that, we hope this approach can be considered as a scalable solution to address national diabetes prevention efforts to target of improvement on diabetes prevalence to not more than 15% by 2025 and serve as a model for applying such services to other chronic diseases.

DETAILED DESCRIPTION:
Digital therapy is a new field that has emerged as the evidence-based treatments from the field of behavioural medicine that are delivered online. It is considered as a scalable method to reach a large number of at-risk population, convenient and accessible. Furthermore, it frees participants from the requirement of travelling to a specific location and more flexible with the time to participate. The aim of this study therefore to determine the feasibility and efficacy of a lifestyle intervention for type 2 diabetes prevention in adults at risk of developing diabetes, an assessor-blinded, parallel-group, randomised controlled trial using the MyDiPP (Malaysia Diabetes Prevention Programme) app. Eligible participants were stratified (age, BMI) and then randomised in a 1:1 ratio to either the 12-month MyDiPP intervention or receive standard health education from primary care providers in the clinic. The study will be conducted in two phases. The first phase will involve preparation of intervention modules, development of intervention mobile app, training and recruitment of participants. The second phase of the study will involve implementation of the intervention, data collection, follow up and data analyses. The study will be conducted in individuals aged 18- to 65-years old, living, working or studying in Kuala Terengganu who is at risk developing diabetes but currently does not have diabetes recruited through online advertisement. The target population is adult residents that lived, worked or studied in Kuala Terengganu who is identified as being at high risk of type 2 diabetes. One hundred participants will be recruited for this study. They will be identified by a two-stage screening process. In the first stage, patients at high risk of type 2 diabetes will be identified via the CDC Diabetes Risk Test that will be distributed via Google Form. The researcher will invite those who scored ≥5 for second stage screening test via the HbA1c test. In the second stage, patients attending a screening for eligibility who have a current HbA1c in the range 38-44 mmol/mol or 5.6-6.2% will be invited to volunteer.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years old
* body mass index (BMI) of ≥23 kg/m2,
* high risk for diabetes (diabetes risk test score ≥5 [22] or HbA1c of 38-44 mmol/mol or 5.6-6.2%
* ownership of a smartphone (Android only) for communication defined as logging on at least once/day to the internet
* being fluent in Malay or English languages and
* had no contradictions to participate in weight management program or physical activity.

Exclusion Criteria:

* clinical history of diabetes or newly diagnosed diabetes at the time of screening where HbA1c level ≥45 mmol/mol or ≥6.3%
* taking oral anti-diabetic agents
* participating in a concurrent weight management program or interventional research protocol
* on a prescribed medical diet, anti-obesity or diabetes therapy within the preceding 4 months
* had clinical history of cardiovascular diseases occurred within the past 6 months
* any form of cancers that require treatment
* dementia or probable Alzheimer's disease
* advanced arthritis
* pregnant or within 6 weeks of having given birth or planning to become pregnant in the next 12 months
* existing liver and renal disease and having hyperthyroidism
* any mental health condition including eating disorder or alcohol/substance use
* other causes which could interfere with participation (for examples physically disabled)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
body weight | 6-months and 12-months
  change of the initial body weight by 5% to 7%

SECONDARY OUTCOMES:
HbA1c level | 6-months and 12-months
  HbA1c level will be tested using A1CNow+ test kit from a finger-stick blood samples collected in a capillary tube according to the manufacturer's procedure guidelines. To measure HbA1c with A1cNow+ test kit, the finger will be cleaned with alcohol swab, allowed to dry and then lanced with sterile lancet to obtain a drop of blood. A 5µl capillary blood sample will be collected and added to the sample dilution buffer. The diluted sample will be mixed and added to the monitoring using transfer pipette. Once the sample was applied, the monitor will begin the analyses. Digital results will be displayed in the display window after 5 minutes. The test result will be recorded for each participant.
physical activity level | 6-months and 12-months
  Physical activity (PA) will be assessed using translated and validated version of short-form International Physical Activity Questionnaire (IPAQ short form). It comprises of seven items that identify frequency and time spent on three specific types of physical activity (walking, moderate intensity activity, and vigorous intensity activity) during the past seven days. The Metabolic Equivalent (MET) values will be measured. The subjects' total physical activity (MET-minutes/week) will be calculated by summing up the walking, moderate and vigorous intensity activity scores. Subjects will be categorised as "active" if they achieved ≥600 MET-minutes/week, "moderately active" if they achieved ≥150 MET-minutes/week and "inactive" if they achieved <150 MET-minutes/week.
dietary intake | 6-months and 12-months
  The dietary intake status of the participants will be assessed from their food diary record from the app and the diary for intervention and control participants respectively. Participants will be asked to record their dietary intake for three days (two weekdays and one weekend) and the average measurement will be taken. A dietary analysis software, Nutritionist Pro Inc. will be used for energy and nutrient analysis.
health-related quality of life | 6-months and 12-months
  HRQoL will be assessed using translated and validated version of SF-36 health survey questionnaire. It comprises of 36 items which measure eight health domains which are physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotion (RE) and mental health (MH). The eight domains will be scored from 0 to 100 indicating worst to best possible health. All the scores will be further summarised into the Physical Component Summary score (PCS) and the Mental Component Summary score (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Sharifah Wajihah Wafa T Syed Saadun Tarek Wafa, PhD, Principal Investigator — Universiti Sultan Zainal Abidin
Locations (1):
- University Sultan Zainal Abidin, Kuala Terengganu, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No